CLINICAL TRIAL: NCT03906175
Title: Whole-body Hyperthermia for Mild to Moderate Depressive Disorder - a Randomized Controlled Tiral
Brief Title: Whole-body Hyperthermia for Mild to Moderate Depressive Disorder
Acronym: HYPE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Holger Cramer, Research Director, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-8439-BO
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Depression, Unipolar
Keywords: Depression; Hyperthermia; Randomized Controlled Trial
MeSH Terms: conditions — Depressive Disorder; Depression; Hyperthermia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-body hyperthermia (Experimental): Whole-body hyperthermia will be applied 2 times during 4 weeks. At week 6, the primary outcome will be assessed. The participants will be reassessed 12 weeks after the start of the treatment with whole-body hyperthermia.
  Interventions: Device: Whole-body hyperthermia
- Wait list (No Intervention): Participants will wait for 6 weeks (primary outcome assessment point). They will then receive the same treatment procedure as the experimental group. They will also be reassessed 12 weeks after the start of the treatment with whole-body hyperthermia.

INTERVENTIONS:
Device: Whole-body hyperthermia — Whole-body hyperthermia will be applied two times during 4 weeks (week 0 and 2 after randomization). The hyperthermia will be applied using Heckel-HT3000 MPIIb.
  Arms: Whole-body hyperthermia

SUMMARY:
The primary aim of this study is to investigate the effectiveness of whole-body hyperthermia in comparison to wait list on depressive symptom severity in patients with mild to moderate depressive disorder currently not under psychotherapeutic or antidepressant drug treatment.

Secondary aims included further quality of life outcomes, immunological parameters, and tolerability/safety of the hyperthermia.

ELIGIBILITY:
Inclusion Criteria:

* Unipolar depression (diagnosed according to the DSM-IV)
* Mild depression: 8-16 points on the HAMD-17 or moderate depression: 17-23 points on the HAMD-17

Exclusion Criteria:

* Current psychotherapy
* Antidepressant drug treatment in the last 4 weeks before study inclusion
* Participants who did not respond to prior antidepressant drug treatment, electroconvulsive therapy, or sleep deprivation (therapy-resistant depression)
* Acute suicidality
* Prior treatment with whole-body hyperthermia
* Contraindications to hyperthermia treatment: acute or feverish infections, severe cardiovascular diseases (e.g. angina pectoris, heart failure, thrombosis, bleeding diathesis), severe gastrointestinal diseases (e.g. renal insufficiency, hepatitis, liver cirrhosis, peptic ulcer), severe neurological diseases (e.g. epilepsy, multiple sclerosis, cerebrovascular malformations or brain tumors), severe endocrine diseases (e.g. hyperthyroidism), or oncological diseases without remission
* Participants taking anti-inflammatory or immunosuppressive drugs
* Participants with severe psychiatric comorbidities (e.g. schizophrenia, schizoaffective disorder, bipolar disorder, dementia, ADHD, obsessive-compulsive disorder, PTSD, alcohol or drug addiction)
* Women during pregnancy and breastfeeding
* Lack of ability to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-06-11 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Depression Severity: clinician-rated | week 6
  Hamilton Rating Scale for Depression (HAMD-17)

SECONDARY OUTCOMES:
Depression Severity: clinician-rated | week 1
  Hamilton Rating Scale for Depression (HAMD-17)
Depression Severity: clinician-rated | week 3
  Hamilton Rating Scale for Depression (HAMD-17)
Depression Severity: clinician-rated | week 12
  Hamilton Rating Scale for Depression (HAMD-17)
Depression Severity: patient-rated | week 1
  Beck Depression Inventory II (BDI-II)
Depression Severity: patient-rated | week 3
  Beck Depression Inventory II (BDI-II)
Depression Severity: patient-rated | week 6
  Beck Depression Inventory II (BDI-II)
Depression Severity: patient-rated | week 12
  Beck Depression Inventory II (BDI-II)
Global improvement: clinician-rated | week 1
  Clinical Global Impression Scale (CGI)
Global improvement: clinician-rated | week 3
  Clinical Global Impression Scale (CGI)
Global improvement: clinician-rated | week 6
  Clinical Global Impression Scale (CGI)
Global Improvement: clinician-rated | week 12
  Clinical Global Impression Scale (CGI)
Global Functioning: clinician-rated | week 1
  Global Assessment of Functioning Scale (GAF)
Global Functioning: clinician-rated | week 3
  Global Assessment of Functioning Scale (GAF)
Global Functioning: clinician-rated | week 6
  Global Assessment of Functioning Scale (GAF)
Global Functioning: clinician-rated | week 12
  Global Assessment of Functioning Scale (GAF)
Fatigue: patient-rated | week 1
  Multidimensional Fatigue Inventory (MFI)
Fatigue: patient-rated | week 3
  Multidimensional Fatigue Inventory (MFI)
Fatigue: patient-rated | week 6
  Multidimensional Fatigue Inventory (MFI)
Fatigue: patient-rated | week 12
  Multidimensional Fatigue Inventory (MFI)
Stress: patient-rated | week 1
  Perceived Stress-Scale (PSS)
Stress: patient-rated | week 3
  Perceived Stress-Scale (PSS)
Stress: patient-rated | week 6
  Perceived Stress-Scale (PSS)
Stress: patient-rated | week 12
  Perceived Stress-Scale (PSS)
Quality of Life: patient-rated | week 1
  Short Form Health Survey (SF-12)
Quality of Life: patient-rated | week 3
  Short Form Health Survey (SF-12)
Quality of Life: patient-rated | week 6
  Short Form Health Survey (SF-12)
Quality of Life: patient-rated | week 12
  Short Form Health Survey (SF-12)
Biomarkers: interleukin 2 | week 1
  IL-2
Biomarkers: interleukin 2 | week 3
  IL-2
Biomarkers: interleukin 2 | week 6
  IL-2
Biomarkers: interleukin 2 | week 12
  IL-2
Biomarkers: interleukin 6 | week 1
  IL-6
Biomarkers: interleukin 6 | week 3
  IL-6
Biomarkers: interleukin 6 | week 6
  IL-6
Biomarkers: interleukin 6 | week 12
  IL-6
Biomarkers: interleukin 10 | week 1
  IL-10
Biomarkers: interleukin 10 | week 3
  IL-10
Biomarkers: interleukin 10 | week 6
  IL-10
Biomarkers: interleukin 10 | week 12
  IL-10
Biomarkers: tumor necrosis factor alpha | week 1
  TNF-alpha
Biomarkers: tumor necrosis factor alpha | week 3
  TNF-alpha
Biomarkers: tumor necrosis factor alpha | week 6
  TNF-alpha
Biomarkers: tumor necrosis factor alpha | week 12
  TNF-alpha
Biomarkers: high-sensitivity C-reactive protein | week 1
  hs-CRP
Biomarkers: high-sensitivity C-reactive protein | week 3
  hs-CRP
Biomarkers: high-sensitivity C-reactive protein | week 6
  hs-CRP
Biomarkers: high-sensitivity C-reactive protein | week 12
  hs-CRP
Biomarkers: soluble intercellular adhesion molecule-1 | week 1
  sICAM-1
Biomarkers: soluble intercellular adhesion molecule-1 | week 3
  sICAM-1
Biomarkers: soluble intercellular adhesion molecule-1 | week 6
  sICAM-1
Biomarkers: soluble intercellular adhesion molecule-1 | week 12
  sICAM-1
Biomarkers: tryptophan | week 1
  tryptophan
Biomarkers: tryptophan | week 3
  tryptophan
Biomarkers: tryptophan | week 6
  tryptophan
Biomarkers: tryptophan | week 12
  tryptophan
Biomarkers: kynurenine | week 1
  kynurenine
Biomarkers: kynurenine | week 3
  kynurenine
Biomarkers: kynurenine | week 6
  kynurenine
Biomarkers: kynurenine | week 12
  kynurenine
Biomarkers: neopterin | week 1
  neopterin
Biomarkers: neopterin | week 3
  neopterin
Biomarkers: neopterin | week 6
  neopterin
Biomarkers: neopterin | week 12
  neopterin
Adverse Events | week 1
  Number of patients with adverse events, total number and type of adverse events
Adverse Events | week 3
  Number of patients with adverse events, total number and type of adverse events
Adverse Events | week 6
  Number of patients with adverse events, total number and type of adverse events
Adverse Events | week 12
  Number of patients with adverse events, total number and type of adverse events

OTHER OUTCOMES:
Treatment Expectations | week -1
  Treatment Credibility Scale (TCS)

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof. MD, Study Director — Center for Integrative Medicine and Health, University Hospital Essen, University of Duisburg-Essen
Locations (1):
- Department of Psychiatry, Psychotherapy and Addiciton Medicine, Evang. Kliniken Essen-Mitte, Essen, Germany

IPD SHARING:
Plan to Share IPD: No